CLINICAL TRIAL: NCT06542562
Title: Accuracy of Fully Guided Versus Half Guided Implant Placement in Patients With Edentulous Maxilla: A Split-mouth Randomized Clinical Trial
Brief Title: Accuracy of Fully Guided Versus Half Guided Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMSA
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2024-07

CONDITIONS: Complete Edentulism
Keywords: implants

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 will undergo fully guided dental implant surgery (Experimental): Group 1 will undergo fully guided dental implant surgery
  Interventions: Procedure: guided implant placement
- Group 2 will undergo half guided dental implant surgery (Experimental): Group 2 will undergo half guided dental implant surgery. Where the implant will be placed after removal of the guide
  Interventions: Procedure: guided implant placement

INTERVENTIONS:
Procedure: guided implant placement — The key difference is that in Group 1, the guide is only used for the drilling sequence, while in Group 2 the guide is used for both the drilling and the actual implant placement.

SUMMARY:
six implants will be placed in edentulous maxilla to rehabilitate patients with implant prosthesis.The primary outcome measure will be the accuracy of implant placement, which will be evaluated using cone-beam computed tomography (CBCT) scans

DETAILED DESCRIPTION:
Study Design:

This will be a Split mouth randomized controlled trial (RCT) study. 16 patients missing teeth in the maxillary (upper) jaw and eligible for dental implant treatment will be recruited.

Interventions will be randomly assigned to the right or the left side of the arch :

Group 1 will undergo fully guided dental implant surgery. Group 2 will undergo partially guided dental implant surgery.

Study Duration:

The total duration of the study is estimated to be 5 months. Recruitment and enrollment of patients: 1 months Dental implant surgery : 3 months Data analysis and manuscript preparation: 1 months

The key steps are:

Recruit 16 eligible patients missing teeth in the maxillary jaw. Randomly assign right or left side of the maxillary arch of patients to either the fully guided or partially guided implant surgery group.

Perform CBCT (cone-beam computed tomography) scans before and after the implant surgery for both groups.

Assess the accuracy of implant placement in both groups using the CBCT data. Conduct statistical analysis to determine if there are any statistically significant differences in implant placement accuracy between the two groups.

Interpret the results and develop recommendations on the optimal guided surgery technique for rehabilitating the edentulous maxilla using dental implants.

The study aims to provide scientific evidence to guide clinicians in selecting the most appropriate guided surgery approach for maxillary implant rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Complete edentulism
* Adequate bone volume to accommodate six standard implant fixtures (3.7 mm diameter and 10 mm length)
* All patients underwent a panoramic X-ray and an oral examination
* Written consent provided prior to participation

Exclusion Criteria:

* Patients with partial edentulism
* Insufficient bone volume for a 3.7 mm diameter and 10 mm length implant fixture
* Local or systemic conditions that could impede dental implant surgery
* Patients who smoke more than five cigarettes per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Rate of Angle Deviation in Implant Placement: Fully Guided vs. Half-Guided Approaches | at the day of implant placement
  Post-surgery, 16 patients will be scanned using the same CBCT machine and exposure settings. Preoperative and postoperative CBCT scans will be imported into the In2Guide™ software, where an overlay of the preoperative plane onto the postoperative scan allowed for precise evaluation of implant positioning. Implant deviations will be measured in three directions: angular deviation, deviation at the coronal platform (entry deviation), and deviation at the apical portion (Figure 2). The software generated coordinates for the necessary calculations, with coronal and apical deviations reported in millimeters and angular deviation in degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- MSA University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alqutaibi AY, Al-Gabri RS, Ibrahim WI, Elawady D. Trueness of fully guided versus partially guided implant placement in edentulous maxillary rehabilitation: a split-mouth randomized clinical trial. BMC Oral Health. 2025 Oct 27;25(1):1680. doi: 10.1186/s12903-025-07073-0. PMID 41146170